CLINICAL TRIAL: NCT00126841
Title: To Assess the Feasibility and Impact of Computed Tomotherapy (CT) and Magnetic Resonance Imaging (MRI) Fusion on Radiation Treatment Planning for Ten Patients With Cancer of the Cervix
Brief Title: Computed Tomotherapy (CT) and Magnetic Resonance Imaging (MRI) Fusion on Radiation Treatment Planning for Patients With Cancer of the Cervix
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: GY-03-0019
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Cervix Cancer
Keywords: radiotherapy planning CT/MR fusion
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: CT and MR fusion

SUMMARY:
Patients with more advanced stages of cervix cancer are treated by radiotherapy. Overall, more than 50% are cured. Approximately half of those patients not cured have current cancer in the irradiated volume. Higher doses of radiation would be expected to cure more patients. To give high doses of radiation safely, the investigators need to know very precisely where the cancer is and then they can use new technology available at the Cross Cancer Institute (tomotherapy) to target the cancer precisely, giving higher doses to the cancerous tissues and lower doses to the non-cancerous tissues.

This study of ten patients with cervical cancer will investigate the added value of MRI scanning on precise tumor definition to facilitate more accurate radiotherapy treatment planning. For this study, patients will be treated in the conventional way with conventional doses. The investigators hope that treatment for future patients will be planned with MRI data and that they will be treated to higher doses of tomotherapy.

DETAILED DESCRIPTION:
Rationale/Background:

For a long time diagnostic imaging has been used in planning radiation treatment for the carcinoma of the cervix, although it is not the essential part of FIGO staging work up. In the past, treatment planning was based on examination under anesthesia (EUA) findings and standard portals were used. Various studies have shown high risks of geographical miss and/or inappropriate tumor coverage (up to >70%) with the use of standard portals, which was related to poor local control. Increasingly, diagnostic/planning CT and MRI imaging are used to plan radiation treatment.

Most patients with invasive carcinoma of the cervix, who are not candidates for radical hysterectomy, are treated by radiotherapy, often with concomitant chemotherapy with a curative intent. Amongst those patients, where cure is not achieved, there are a significant proportion who fail first or only in the pelvis. Higher doses of radiation would be expected to reduce this risk. With conventional radiotherapy, higher doses of radiation result in a higher rate of complications. New technology available at the Cross Cancer Institute (tomotherapy + intensity modulated radiation therapy [IMRT]) would be expected to permit higher doses of radiation to be delivered but avoid the increased risk of complications. Accurate definition of clinical target volume, composed of the cervix, uterus, gross primary tumor and the regional lymphatic drainage is required for accurate treatment planning. The MRI imaging is expected to be valuable in this regard. Demonstrating this is the immediate aim of this study. The investigators' long term aim will be to replace conventional external beam radiotherapy with helical tomotherapy. They expect to be able to apply increasing doses of radiation to the GTV + CTV and monitor short-term treatment effects with biological imaging, principally magnetic resonance spectroscopy (MRS). Eventually the investigators hope to be able to individualize radiation doses based in part on biological imaging, before and during treatment.

In their center the investigators routinely perform diagnostic and planning CT scans of almost all Ca. cervix patients before radiation treatment planning. This study will involve one additional MRI scan of the pelvis, which will take about 30 minutes to perform; this process has potential benefit in the treatment planning.

Studies comparing imaging modalities for diagnostic accuracy:

There are studies in which CT and MRI scans were performed preoperatively and results were compared with surgical-pathological outcome to confirm their diagnostic accuracy in terms of tumor detection, parametrial invasion, lymph node status and adjacent organ involvement. MRI was consistently reported to be more accurate than CT scan in terms of tumor delineation and normal organ localization. This is also true for a meta-analysis of 17 eligible studies.

Studies Comparing Imaging Modalities for Treatment Planning:

Not surprisingly CT planning was shown to be superior over standard field technique for external beam radiation therapy (EBRT) and brachytherapy planning for ca cervix patients. There was less chance of geographical miss by using an imaging modality for planning. Studies comparing MRI and CT for treatment planning showed that MRI led to significant changes in field borders.

Image Fusion:

Harms W et al from Germany studied the fusion of CT and MRI images from sixteen patients who were treated by interstitial (n=12) and endocavitary (n=4) brachytherapy for recurrent cervix, head and neck, sarcoma and vulva carcinoma. They compared conventional 3D-brachytherapy planning based on CT-information alone to brachytherapy planning based on fused CT and MRI data. They measured the accuracy of image fusion using predefined corresponding landmarks in the CT and MRI data. They found that an automated algorithm was robust and reliable (mean registration error 1.8 mm, range 0.8-4.1 mm, SD 0.9 mm); tumor visualization was difficult using CT alone; and brachytherapy treatment planning based on fused CT and MRI data enabled better definition of target volume and critical structures as compared to treatment planning based on CT alone.

Patients and Methods:

Ten patients with a histological diagnosis of cervix carcinoma who are to receive treatment at the Cross Cancer Institute will be enrolled in this fusion study. They will go through the usual investigations prior to treatment planning, including CT imaging. In addition, patients will have an MRI of the pelvis which takes approximately about 30 minutes.

CT and MRI imaging will be fused using fusion software. Treatment planning for standard four field box technique and tomotherapy will be done on CT images as usual and subsequently on fused images. Tumor coverage and normal organ doses will be recorded and compared. Tumor control probabilities and normal tissue complication probabilities will be calculated for the different plans to facilitate objective comparisons.

Conclusion:

Most patients with invasive carcinoma of the cervix, who are not candidates for a radical hysterectomy, are often treated by concomitant chemo-radiation with a curative intent. Patients who cannot achieve a cure with this treatment fail first or only in the pelvis. The higher doses of radiation would be expected to reduce this risk, which cannot be achieved with conventional radiotherapy due to higher rates of complications. Tomotherapy based treatment planning would be expected to obtain higher doses of radiation to be delivered but avoid the measured risk of complications. More accurate definition of clinical target volume, composed of the cervix, uterus, gross primary tumor and the regional lymphatic drainage is required for accurate treatment planning. Currently the investigators are planning on the basis of CT scan only in their center; MRI scan is consistently shown to be superior over CT for treatment. Fusing MRI and CT images are expected to delineate structures more accurately compared to CT alone and therefore will be valuable in accurate treatment planning to deliver higher doses to CTV without increasing treatment related complications.

Objectives:

1. To assess the feasibility of image fusion between MRI and CT for radiotherapy (RT) planning in Ca. Cervix
2. To determine the added value of fused MRI and CT over CT alone for RT planning.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer undergoing primary radiotherapy

Exclusion Criteria:

* Stage 1B
* Patient refusal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 10
Dates: Start 2004-11; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearcey, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Subak LL, Hricak H, Powell CB, Azizi L, Stern JL. Cervical carcinoma: computed tomography and magnetic resonance imaging for preoperative staging. Obstet Gynecol. 1995 Jul;86(1):43-50. doi: 10.1016/0029-7844(95)00109-5. PMID 7784021
- [Background] Ozsarlak O, Tjalma W, Schepens E, Corthouts B, Op de Beeck B, Van Marck E, Parizel PM, De Schepper AM. The correlation of preoperative CT, MR imaging, and clinical staging (FIGO) with histopathology findings in primary cervical carcinoma. Eur Radiol. 2003 Oct;13(10):2338-45. doi: 10.1007/s00330-003-1928-2. Epub 2003 Jun 12. PMID 12802611
- [Background] Kim SH, Choi BI, Han JK, Kim HD, Lee HP, Kang SB, Lee JY, Han MC. Preoperative staging of uterine cervical carcinoma: comparison of CT and MRI in 99 patients. J Comput Assist Tomogr. 1993 Jul-Aug;17(4):633-40. doi: 10.1097/00004728-199307000-00022. PMID 8331236
- [Background] Ho CM, Chien TY, Jeng CM, Tsang YM, Shih BY, Chang SC. Staging of cervical cancer: comparison between magnetic resonance imaging, computed tomography and pelvic examination under anesthesia. J Formos Med Assoc. 1992 Oct;91(10):982-90. PMID 1362678
- [Background] Bipat S, Glas AS, van der Velden J, Zwinderman AH, Bossuyt PM, Stoker J. Computed tomography and magnetic resonance imaging in staging of uterine cervical carcinoma: a systematic review. Gynecol Oncol. 2003 Oct;91(1):59-66. doi: 10.1016/s0090-8258(03)00409-8. PMID 14529663
- [Background] Scheidler J, Hricak H, Yu KK, Subak L, Segal MR. Radiological evaluation of lymph node metastases in patients with cervical cancer. A meta-analysis. JAMA. 1997 Oct 1;278(13):1096-101. PMID 9315770
- [Background] Knocke TH, Pokrajac B, Fellner C, Potter R. [A comparison of CT-supported 3D planning with simulator planning in the pelvic irradiation of primary cervical carcinoma]. Strahlenther Onkol. 1999 Feb;175(2):68-73. doi: 10.1007/BF02753845. German. PMID 10065141
- [Background] Wachter-Gerstner N, Wachter S, Reinstadler E, Fellner C, Knocke TH, Potter R. The impact of sectional imaging on dose escalation in endocavitary HDR-brachytherapy of cervical cancer: results of a prospective comparative trial. Radiother Oncol. 2003 Jul;68(1):51-9. doi: 10.1016/s0167-8140(03)00083-5. PMID 12885452
- [Background] Krempien RC, Daeuber S, Hensley FW, Wannenmacher M, Harms W. Image fusion of CT and MRI data enables improved target volume definition in 3D-brachytherapy treatment planning. Brachytherapy. 2003;2(3):164-71. doi: 10.1016/S1538-4721(03)00133-8. PMID 15062139